CLINICAL TRIAL: NCT01545128
Title: A Retrospective Case-control Study Comparing the Direrct Healthcare Costs of Conventionally Managed COPD Patients With Those Who Have Completed a Pulmonary Rehabilitation Programme
Brief Title: Impact of Pulmonary Rehabilitation on Direct Healthcare Costs in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Principal Investigator, Indranil Chakravorty, Consultant Physician, East and North Hertfordshire NHS Trust
Other Study IDs: 07/H0311/87
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: COPD
Keywords: COPD; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study the direct cost of illness study of COPD patients who participated in a Pulmonary rehabilitation program for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* COPD

Exclusion Criteria:

* None

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: copd
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-01; Study Completion 2010-01 (Actual)